CLINICAL TRIAL: NCT05015309
Title: A Phase I, Open-Label Study to Determine Safety, Tolerability, Pharmacokinetics (PK) and Preliminary Efficacy of SH3765 Tablet in Patients With Advanced Malignant Tumor
Brief Title: A Study to Investigate Safety and Tolerability of SH3765 Tablet in Patients With Advanced Malignant Tumor
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanjing Sanhome Pharmaceutical, Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SHC039-I-01
Record Dates: First submitted 2021-08-18; First posted 2021-08-20 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Advanced Malignant Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SH3765 tablet (Experimental): Daily oral administration of SH3765 tablet
  Interventions: Drug: SH3765 tablet

INTERVENTIONS:
Drug: SH3765 tablet — Starting dose 2.5mg, oral administered once daily. If tolerated subsequent cohorts will test increasing doses (5mg, 10mg, 15mg, 20mg, 25mg, 30mg) of SH3765.

SUMMARY:
The primary objective is to determine the safety and tolerability of SH3765 in subjects with advanced malignant tumor by determining the maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D). The second objective is to evaluate the PK profile and preliminary efficacy of SH3765 in subjects with advanced malignant tumor.

DETAILED DESCRIPTION:
This is a Phase I, open-label, multicenter, multidose, two-part study to assess the safety, tolerability, PK and preliminary efficacy of SH3765, a protein arginine methyltransferase 5 (PRMT5) inhibitor, in subjects with advanced malignant tumor including but not limited to solid tumor and non-Hodgkin lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Patients must have a histologically or cytologically confirmed diagnosis of relapsed or refractory solid tumors or non-Hodgkin lymphomas (NHLs), with the following criteria specific to each tumor type:

   For solid tumors: Patients must have advanced triple-negative breast cancer (TNBC), non-small cell lung cancer (NSCLC), adenoid cystic carcinoma (ACC), prostate cancer (PC), or head and neck squamous cell carcinoma (HNSCC). The malignancy must be relapsed or refractory after at least 1 prior line of anti-tumor therapy, and for which there are no available standard of care therapy or therapies known to provide clinical benefit; For NHLs: Patients must have mantle cell lymphoma (MCL), or non-germinal center B-cell-like (non-GCB) subtypes of diffuse large B-cell lymphoma (DLBCL) (both de novo and transformed non-GCB DLBCL are allowed). The malignancy must be relapsed or refractory after at least 2 prior lines of anti-tumor therapy, and for which there are no available standard of care therapy or therapies known to provide clinical benefit. The patients who require urgent cytoreductive therapy will be excluded, unless the patient has no remaining treatment choice with potential benefits.
3. Patients must provide archival tumor tissue, if available, from the most recent biopsy, or are able to undergo a tumor biopsy during screening;
4. At least one evaluable or measurable tumor lesion;
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1;
6. Life expectancy ≥3 months;
7. Adequate hematological and biological function, confirmed by the following laboratory values (Have not received blood transfusion or hematopoietic stimulating factor treatment within 14 days):APTT ≤1.0×ULN; Total bilirubin (TBIL) ≤1.5×ULN if no demonstrable liver lesion(s) (primary or metastases) or ≤3×ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinemia) or liver lesion(s); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN if no demonstrable liver lesion(s) (primary or metastases) or ≤5×ULN in the presence of liver lesion(s); Creatinine clearance ≥50mL/min (Calculated according to Cockcroft-Gault formula); Left ventricular ejection fraction (LVEF) ≥50%; QT interval corrected using Fridericia's method (QTcF)<470 msec; For advanced solid tumors patients: ANC ≥1.5×109/L, PLT ≥100×109/L, Hemoglobin (Hb) ≥90 g/L; For advanced non-Hodgkin lymphoma patients: ANC ≥ 1.0×109/L, PLT ≥ 80×109/L, Hemoglobin (Hb) ≥80 g/L;
8. Women of child bearing potential must agree to use a reliable form of contraception during the study treatment period and for at least 180 days following the last dose of study drug, and 3 days before treatment the pregnancy tests are negative. Men must agree to the use of male contraception during the study treatment period and for at least 180 days after the last dose of study drug;
9. Not using any other investigational drugs within 30 days before the study drugs administration;
10. Be informed of the trial before the start of the trial, and voluntarily sign the name and date on the informed consent form.

Exclusion Criteria:

1. Prior treatment with PRMT5 inhibitors;
2. Anticancer treatment including radiation therapy, chemotherapy, hormonal therapy, molecular targeted therapy, or immunotherapy within 3 weeks before the first dose of SH3765 (use of mitomycin or nitrosoureas within 6 weeks before the first dose; use of oral fluorouracil, such as tegafur and capecitabine, within 2 weeks before the first dose; use herbal medicine with anti-tumor indications within 2 weeks before the first dose);
3. Evidence of central nervous system (CNS) metastases;
4. Evidence of any severe or uncontrolled systemic diseases, including uncontrolled hypertension, active bleeding diatheses, uncontrolled pleural effusion and ascites, uncontrolled diabetes, non-infectious pneumonia, or any other severe cardiovascular, respiratory, nervous and mental diseases;
5. Have severe cardiac disease:NYHA class ≥grade II heart failure; arrhythmia requiring medical treatment; myocardial infarction or unstable angina pectoris within 6 months; currently taking known QT extension drugs those who cannot stop the drug for at least 5 half-lives before starting the study drug treatment；
6. Patients who have active infection within 1 week before the first administration and need systematic anti-infection treatment;
7. Active infection with hepatitis B virus (HBV), hepatitis C virus (HCV) or human immunodeficiency virus (HIV). Patients with HBsAg positive but HBV-DNA negative, or with HCV antibody positive but HCV-RNA negative, or with HIV antibody positive but HIV-RNA negative and CD4+ T cell count normal will be inclusive;
8. Patients who received systemic glucocorticoids (prednisone >10 mg/ day or equivalent dose of the same drug) or other immunosuppressive therapy within 14 days before the first administration; except for topical, ocular, intra-articular, intranasal, and inhaled glucocorticoids; short-term use of glucocorticoids for prophylactic treatment (e.g., prevention of contrast agent allergy);
9. The patient is currently using (or cannot stop at least 1 week prior to the first administration of the study drug) a drug known to be a strong inhibitor or inducer of CYP3A4 and inhibitor of P-gp;
10. Patients who received granulocyte colony stimulating factor (G-CSF) or blood transfusion therapy within 7 days before the hematologic examination at the screening stage;
11. Autologous hematopoietic stem cell transplantation was performed within 90 days prior to the start of the study;
12. Previous recipients of allogeneic hematopoietic stem cell transplantation or organ transplantation;
13. According to CTCAE 5.0, adverse reactions from previous anti-tumor therapy have not yet returned to ≤ grade 1 (except for toxicities which are judged by researchers to be safe, such as hair loss)；
14. Had major organ surgery (excluding puncture biopsy) or had significant trauma within 4 weeks before the first administration, or needed to undergo surgery during the trial period;
15. Uncontrolled nausea and vomiting, chronic gastrointestinal disease, inability to swallow pharmaceutical preparations, extensive enterectomy and possible impairment of adequate absorption of study drugs;
16. According to CTCAE 5.0, experiencing any CTCAE grade 3 or 4 gastrointestinal bleeding in the 3 months prior to enrollment;
17. Allergic to the similar drug or its excipients;
18. Lactating women;
19. The investigator determined that the patient should not participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Within the first 28 days of consecutive treatment
  DLT is defined as an adverse event that meets protocol defined DLT criteria occurring from the first dose to the end of cycle 1 of multiple doses, except those unequivocally due to the underlying malignancy or an extraneous cause.
Maximum tolerated dose (MTD) | Within the first 28 days of consecutive treatment
  MTD was defined as the highest dose at which DLT occurred in less than one-third of subjects during the DLT observation period.

SECONDARY OUTCOMES:
Cmax | 4 weeks
  Highest observed plasma concentration of SH3765
Tmax | 4 weeks
  Time of highest observed plasma concentration of SH3765
T1/2 | 4 weeks
  Elimination half-life of SH3765
Area Under the Curve (AUC) | 4 weeks
  Area under the plasma concentration time curve of SH3765
Mean Residence Time (MRT) | 4 weeks
  The average residence time in body of SH3765
Overall Response Rate (ORR) | up to 12 months
Progression-free survival (PFS) | up to 12 months
Disease control rates (DCR) | up to 12 months
Duration of response (DOR) | up to 12 months
Lymph node response rate (LNR) | up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China